CLINICAL TRIAL: NCT02069704
Title: Open Label Randomized Bioequivalence Study to Evaluate the Pharmacokinetic and Safety Profile of Bevacizumab Biosimilar (BEVZ92) vs Bevacizumab (AVASTIN®), Both With FOLFOX or FOLFIRI, in First-line Treatment for mCRC Patients
Brief Title: Bioequivalence Study Bevacizumab Biosimilar (BEVZ92) Versus Bevacizumab (AVASTIN®) in First-line Treatment mCRC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Collaborators: Laboratorio Elea Phoenix S.A. (Industry); Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEVZ92-A-01-13; BEVZ92-A-01-13 (Registry Identifier: BEVZ92-A-01-13)
Record Dates: First submitted 2014-02-14; First posted 2014-02-24 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: colorectal cancer; metastatic; first-line treatment; comparability
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — BEVZ92; Fluorouracil; Oxaliplatin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab biosimilar (BEVZ92) (Experimental): Bevacizumab 25 mg/mL (strength: 100 mg/4 mL).
  Interventions: Drug: Bevacizumab biosimilar (BEVZ92)
- Avastin® (bevacizumab, ref. product) (Active Comparator): Bevacizumab 25mg/ml (strength: 100mg/4ml)
  Interventions: Drug: Avastin® (bevacizumab, reference product)

INTERVENTIONS:
Drug: Bevacizumab biosimilar (BEVZ92) — Active ingredient Bevacizumab 25 mg/mL (strength = 100 mg/4 mL). 30-minute* IV infusion (5 mg/kg) every 2 weeks, prior to chemotherapy (Folfox any or Folfiri).
  FOLFIRI = Folinic Acid + Fluorouracil + Irinotecan FOLFOX = Folinic Acid + Fluorouracil + Oxaliplatin Treatment will continue until disease progression, unacceptable toxicity, patient withdraws consent or death (whichever occurs first).
  *The first infusion will be given over 90 minutes. If it is well tolerated, the second infusion can be given over 60 minutes. If it is well tolerated, subsequent infusions can be given over 30 minutes.
  The FOLFOX (any) or FOLFIRI regimen will be chosen as per investigator's criteria based on the hospital standard of care.
  Other Names: FOLFOX = Folinic acid + Fluorouracil + Oxaliplatin; FOLFIRI = Folinic acid + Fluorouracil + Irinotecan
  Arms: Bevacizumab biosimilar (BEVZ92)
Drug: Avastin® (bevacizumab, reference product) — Active ingredient: Bevacizumab 25 mg/mL (strength: 100 mg/4 mL). 30-minute* IV infusion (5 mg/kg) every 2 weeks, prior to administration of chemotherapy. Treatment will continue until disease progression, unacceptable toxicity, patient withdraws consent or death (whichever occurs first).
  *The first infusion will be given over 90 minutes. If the first infusion is well tolerated, the second infusion can be given over 60 minutes. If this infusion is well tolerated, subsequent infusions can be given over 30 minutes.
  The FOLFOX (any) or FOLFIRI regimen will be chosen as per investigator's criteria based on the hospital standard of care.
  Other Names: FOLFOX = Folinic acid + Fluorouracil + Oxaliplatin; FOLFIRI = Folinic acid + Fluorouracil + Irinotecan
  Arms: Avastin® (bevacizumab, ref. product)

SUMMARY:
This is a multicenter, open label, randomized bioequivalence study of BEVZ92 (bevacizumab biosimilar) and Avastin® with 2 parallel arms to compare the pharmacokinetic (PK) profile of BEVZ92 and Avastin® in combination with FOLFOX (any) or FOLFIRI chemotherapy.

FOLFOX (any) or FOLFIRI will be chosen as per investigator criteria based on the hospital standard of care.

DETAILED DESCRIPTION:
Planned enrolment duration: 12 months. Pre-treatment period (included in enrolment period): 1 month. Treatment period: Patients will continue treatment until disease progression or unacceptable toxicity, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must not have had prior chemotherapy for advanced or metastatic disease. Patients could have received adjuvant chemotherapy or adjuvant chemo-radiotherapy.
2. Patient with mCRC for whom bio-chemotherapy is indicated.
3. Patients must have at least one measurable non-irradiated site of disease according to RECIST (version 1.1) criteria. If the patient has had previous irradiation of the marker lesion(s), there must be evidence of progression since the radiation.
4. Minimum of 4 weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Adequate bone marrow function
7. Adequate liver function defined within specific parameters
8. Adequate renal function defined within specific parameters
9. Adequate coagulation parameters defined within specific parameters
10. Negative pregnancy test for females of a childbearing potential.
11. Use of an effective form of contraception during the study (for subjects of childbearing potential and their partners).
12. Life expectation ≥ 3 months

Exclusion Criteria:

1. Prior treatment for advanced or metastatic colorectal cancer.
2. Prior treatment with an anti-angiogenesis agent, in either the neoadjuvant or adjuvant setting.
3. Concurrent use of investigational anti-neoplastic agents (including up to 4 weeks prior to enrolment).
4. History of any other malignancy unless the malignancy is in complete remission and the patient has been off all therapy for that malignancy for at least 5 years.
5. Chronic treatment with systemic steroids or other immunosuppressive agents; topical or inhaled corticosteroids are allowed.
6. Scheduled immunization with attenuated live vaccines during study period or within 1 week prior to study entry.
7. Uncontrolled brain or lepto-meningeal metastases, including patients who continue to require glucocorticoids for brain or lepto-meningeal metastases.
8. Patients with active bleeding or history of bleeding diathesis on oral anti-vitamin K medication (except low dose coumadin) within the past 6 month prior to randomization or coagulopathy.
9. Patients with history of cerebral vascular accident, transient ischemic attack, or subarachnoid haemorrhage within the past 6 month prior to randomization.
10. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
11. Patients with serious non-healing wound, ulcer, bone fracture, or with a major surgical procedure, or significant traumatic injury within 4 weeks prior to randomization
12. Patients with clinical symptoms or signs of gastrointestinal obstruction that require parenteral hydration and/or nutrition.
13. Patients with history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months prior to randomization.
14. Patients with history of hypersensitivity to any of the study drugs or ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Argentina (2):
  - Hospital de Gastroenterologia "Dr. Carlos Bonorino Udaondo", Buenos Aires
  - Instituto Oncológico de Rosario, Rosario
- Brazil (6):
  - Fundaçáo Pio XII - Hospital do Cancer de Barretos, Barretos
  - Hospital Caridade, Ijuí
  - Hospital Sao Lucas da Pucrs, Porto Alegre
  - Centro de Pesquisa do Instituto Brasileiro de Controle do Câncer - IBCC, São Paulo
  - Hosp. A.C Camargo, São Paulo
  - Instituto do Cancer del estado de S. Paulo (ICEPS ), São Paulo
- India (6):
  - M S Patel Cancer Centre- Shree Krishna Hospital, Karamsad, Gujarat
  - Sri Ramachandra Hospital, Chennai
  - Tata Hospital, Mumbai
  - Central India Canter Research Institute, Nagpur
  - Curie Manavta Cancer Center, Nashik
  - Regional Cancer Center & Medical College, Thiruvananthapuram
- Centro Oncológico Clara Campal, Madrid, Spain
- Ukraine (3):
  - Dnipropetrovsk City Multiple-discipline Clinical Hospital №4, Dnipropetrovsk
  - Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Danylo Halytskiy Lviv National Medical University, Lviv

REFERENCES:
- [Derived] Romera A, Peredpaya S, Shparyk Y, Bondarenko I, Mendonca Bariani G, Abdalla KC, Roca E, Franke F, Melo Cruz F, Ramesh A, Ostwal V, Shah P, Rahuman SA, Paravisini A, Huerga C, Del Campo Garcia A, Millan S. Bevacizumab biosimilar BEVZ92 versus reference bevacizumab in combination with FOLFOX or FOLFIRI as first-line treatment for metastatic colorectal cancer: a multicentre, open-label, randomised controlled trial. Lancet Gastroenterol Hepatol. 2018 Dec;3(12):845-855. doi: 10.1016/S2468-1253(18)30269-3. Epub 2018 Sep 24. PMID 30262136

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab Biosimilar (BEVZ92): Bevacizumab biosimilar (BEVZ92): Bevacizumab biosimilar (BEVZ92), Active ingredient Bevacizumab 25 mg/mL (strength = 100mg/mL). 30-minute* IV infusion (5 mg/kg) every 2 weeks, prior to chemotherapy (Folfox any or Folfiri).
- Avastin® (Bevacizumab, Ref. Product): Avastin® (bevacizumab, reference product): Avastin® (bevacizumab, reference product).
  Active ingredient: Bevacizumab 25 mg/mL (strength: 100 mg/4 mL). 30-minute* IV infusion (5 mg/kg) every 2 weeks, prior to administration of chemotherapy (Folfox any or Folfiri).
Period: Overall Study
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product)
Started | 69 (Two patients were randomized but they did not received study treatment) | 71
Completed | 69 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product) | Total
Number analyzed (Participants) | 69 | 71 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (12.9) | 56.7 (11.6) | 56.5 (12.2)
Age, Customized [Count of Participants; unit: Participants]
  Aged: < 65 years | 49 | 51 | 100
  Aged: >= 65 years | 20 | 20 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 39 | 39 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 50 | 55 | 105
  Race: Asian | 14 | 12 | 26
  Race: Black | 2 | 3 | 5
  Race: Other | 3 | 1 | 4
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — Describes a patient's ability to selfcare, daily activity and physical ability. Grades:
  0. Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; about >50% of waking hours.
  3. Capable of only limited selfcare; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair.
  5. Dead.
  Participants
    0 | 7 | 18 | 25
    1 | 57 | 43 | 100
    2 | 5 | 10 | 15
Tumor, lymph Nodes and Metastases (TNM) stage [Count of Participants; unit: Participants] — The TNM Classification of Malignant Tumors describes the stage of a solid tumor according to:
  1. Primary tumour (T)- the size and whether it has invaded nearby tissue, from 0 [no evidence of tumor] to 4 [the highest size and/or extension]
  2. Lymph nodes (N) describes nearby (regional) lymph nodes that are involved, from 0 [no evidence of tumor] to 3 [high extension and numerous lymph nodes],
  3. Metastasis (M) describes distant metastasis, from 0 (no metastases) to 1 (yes). Stage IVa: Any T, Any N, M1a (to the other lung); Stage IVb: Any T, Any N, M1b or M1c ( outside of the chest)
  Participants
    IVa | 30 | 32 | 62
    IVb | 38 | 38 | 76
    missing | 1 | 1 | 2
Months since diagnosis of metastatic colorectal cancer [Mean (Standard Deviation); unit: months] — Population: Missing data for two patients in each treatment arm
  months
    number analyzed (Participants) | 67 | 69 | 136
    (all) | 13.0 (14.7) | 13.0 (17.5) | 13.0 (16.1)
Number of target lesions [Count of Participants; unit: Participants]
  1 | 9 | 11 | 20
  2 | 29 | 31 | 60
  >=3 | 31 | 29 | 60
Extent of disease [Count of Participants; unit: Participants]
  Liver disease only | 7 | 5 | 12
  Other | 62 | 66 | 128
Previous treatment [Number; unit: participants]
  Surgery | 55 | 53 | 108
  Radiotherapy | 14 | 15 | 29
  Chemotherapy | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-versus-time Curve (AUC) at Cycle 1 (AUC0-336h) of BEVZ92 and Avastin®
Description: To compare the pharmacokinetic (PK) profile of BEVZ92 and Avastin®, both administered in combination with FOLFOX (any) or FOLFIRI, by means of comparing the truncated AUC calculated from start of the first infusion until start of the second infusion (i.e. at Cycle 1; AUC0-336h)
  For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) of the ratio of a log-transformed exposure measure (AUC) falls completely within the range 80-125%.
Time Frame: AUC0-336 hrs: 0 to 336 hours after start of the first infusion
Population: Overall number of participants Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Groups:
- Bevacizumab Biosimilar (BEVZ92): Bevacizumab proposed biosimilar (BEVZ92)
- Avastin® (Bevacizumab, Ref. Product).: Avastin® (bevacizumab, reference product).
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 55 | 61
ng.h/mL | 16500000 (30.7) | 16600000 (31.8)
Statistical Analysis 1: Comparison: Bevacizumab Biosimilar (BEVZ92) vs Avastin® (Bevacizumab, Ref. Product); Based on previously published PK data for reference bevacizumab in metastatic colorectal cancer, we assumed a conservative inter-participant coefficient of variation for AUC of around 35%. A sample size of 51 patients in each treatment arm could show bioequivalence with a nominal power of 90% and an α of 0·05, if the 90% CIs for the ratio of BEVZ92 to reference bevacizumab of the geometric means for AUC0-336h and AUCss were within the acceptance interval of 80%-125%; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (AUC) falls completely within the range 80%-125%; ratio BEVZ92 to Avastin = 99.4, 90% CI 2-sided [90.5 to 109.0] — For the ratio: BEVZ92 represents the numerator and reference bevacizumab the denominator

2. Primary Outcome: AUC at Steady State (AUCss) of BEVZ92 and Avastin®
Description: To compare the PK profile of BEVZ92 and Avastin®, both administered in combination with FOLFOX (any) or FOLFIRI, by means of comparing the truncated area under the concentration-versus-time curve calculated over a dosage interval at steady state (i.e. at Cycle 7; AUCss).
  For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (AUC) falls completely within the range 80-125%.
Time Frame: AUCss: 0 to 336 hours after the administration of Cycle 7 infusion (Week 13).
Population: In the Avastin arm there were 3 missing samples at the timepoint required for the specific PK parameters within Cycle 7.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Groups:
- Bevacizumab Biosimilar (BEVZ92): Bevacizumab proposed biosimilar (BEVZ92):
  Active ingredient Bevacizumab 25 mg/mL (strength = 100mg/mL). 30-minute* IV infusion (5 mg/kg) every 2 weeks, prior to chemotherapy (Folfox any or Folfiri).
- Avastin® (Bevacizumab, Ref. Product).: Bevacizumab reference product: Active ingredient Bevacizumab 25 mg/mL (strength = 100mg/mL). 30-minute* IV infusion (5 mg/kg) every 2 weeks, prior to chemotherapy (Folfox any or Folfiri).
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 55 | 58
ng.h/mL | 35900000 (34.8) | 35700000 (36.6)
Statistical Analysis 1: Comparison: Bevacizumab Biosimilar (BEVZ92) vs Avastin® (Bevacizumab, Ref. Product); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ratio BEVZ92 to Avastin = 100.0, 90% CI 2-sided [90.2 to 112.0]

3. Secondary Outcome: Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) Reported With BEVZ92 and Avastin®
Description: Compare the safety profile by means of the frequency and severity of TEAEs and SAEs reported in each treatment arm.
Time Frame: From first study dose and up to 30 days after the end of study treatment for each patient, for an average of 11 months
Population: All patients receiving at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product)
Number analyzed (Participants) | 69 | 71
participants
  Any TEAE (any causality) | 66 | 71
  Any grade>=3 TEAE | 44 | 49
  Any TEAE leading to discontinuation | 13 | 6
  Any treatment-related TEAE | 63 | 70
  Any grade >=3 treatment-related TEAE | 63 | 70
  Any serious TEAE | 19 | 21
  Any bleeding event | 14 | 19

4. Secondary Outcome: Anti-Drug Antibody (ADA) of BEVZ92 and Avastin®
Description: Immunogenicity profile by means of measurement of ADA developed de novo (seroconversion) after cycle 5, cycle 8, and 12 months after first drug administration (pre-dose).
Time Frame: At baseline, and on Day 1 (pre-dose) of Cycles: 1, 5 and 8, and 12 months after first drug administration
Population: All patients receiving at least one dose of study medication.
Measure: Number; unit: participants
Groups:
- Avastin® (Bevacizumab, Ref. Product): Bevacizumab 25mg/ml (strength: 100mg/4ml)
  Avastin® (bevacizumab, reference product): Avastin® (bevacizumab, reference product).
  Active ingredient: Bevacizumab 25 mg/mL (strength: 100 mg/4 mL). 30-minute* IV infusion (5 mg/kg) every 2 weeks, prior to administration of chemotherapy (Folfox any or Folfiri).
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product)
Number analyzed (Participants) | 69 | 71
participants
  Seroconversion | 2 | 0
  No seroconversion | 67 | 71

5. Secondary Outcome: Objective Response Rate (ORR) of BEVZ92 and Avastin®
Description: To compare efficacy in terms of ORR between arms. Clinical and radiological tumor assessments were performed according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 using computed tomography (CT) or magnetic resonance imaging (MRI) scans.
  Objective response (OR) is defined as a best overall response of partial response (PR) or complete response (CR) as defined by RECIST v1.1. All participants who did not meet the criteria for CR or PR by the end of the study were considered non-responders.
Time Frame: Every four weeks. Up to 48 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product)
Number analyzed (Participants) | 71 | 71
Participants
  ORR (CR+PR) | 35 | 40
  Stable disease | 27 | 25
  Progressive disease | 4 | 2
  unevaluable | 5 | 4

6. Secondary Outcome: Cmax,sd of BEVZ92 and Avastin®
Description: Secondary PK endpoints included the Cmax calculated at Cycle 1 (Cmax,sd )
Time Frame: Cmax, sd: 0 to 336 hours after start of the first infusion.
Population: Overall number of participants Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 55 | 61
ng/mL | 120000 (30) | 123000 (27.2)

7. Secondary Outcome: Progression-free Survival (PFS) of BEVZ92 and Avastin®
Description: Compare PFS between the randomized treatment arms. Progression-free survival (PFS) was defined as the time from the randomization date to the date of disease progression using RECIST v1.1, or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions plus 5 mm absolute increase, and/or unequivocal progression of known non-target lesion, and/or the appearance of new lesions".
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 weeks.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product)
Number analyzed (Participants) | 71 | 71
months | 10.8 [7.4 to 11.5] | 11.1 [8.6 to 12.8]

8. Secondary Outcome: Cmax,ss of BEVZ92 and Avastin®
Description: Secondary PK endpoints included the Cmax calculated at Cycle 7 (Cmax, ss )
Time Frame: Cmax, ss: 0 to 336 hours post-dose after the administration of Cycle 7 infusion (Week 13)
Population: In the Avastin arm there were 3 missing samples at the timepoint required for the specific PK parameter within Cycle 7.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 55 | 58
ng/mL | 195000 (29.5) | 200000 (30.7)

9. Secondary Outcome: Ctrough,sd of BEVZ92 and Avastin®
Description: Secondary PK endpoints included the Ctrough calculated at Cycle 1 (Ctrough,sd )
Time Frame: Ctrough, sd: 0 to 336 hours after start of the first infusion.
Population: In the Avastin arm there was 1 missing samples at the timepoint required for the specific PK parameter within Cycle 1.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 55 | 60
ng/mL | 344 (12.5) | 349 (13.7)

10. Secondary Outcome: Ctrough,ss of BEVZ92 and Avastin®
Description: Secondary PK endpoints included the Ctrough calculated at Cycle 7 (Ctrough,ss)
Time Frame: Ctrough, ss: 0 to 336 hours after the administration of the Cycle 7 infusion.
Population: There were 4 missing samples (1 in the BEVZ92 and 3 in the Avastin arm) at the timepoint required for the specific PK parameter within Cycle 7.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 54 | 58
ng/mL | 69600 (52.1) | 69300 (50.5)

11. Secondary Outcome: Elimination Half-life (t1/2) of BEVZ92 and Avastin®
Description: Secondary PK endpoints included the t1/2 calculated at Cycle 7
Time Frame: t1/2: 0 to 336 hours after the administration of the Cycle 7 infusion.
Population: In the Avastin arm there were several missing samples at the timepoint required for the specific PK parameter
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 49 | 52
h | 294 (33.3) | 289 (32.8)

12. Secondary Outcome: Elimination Rate Constant (Kel) of BEVZ92 and Avastin®
Description: Secondary PK endpoints included the Kel calculated at Cycle 7 (Ctrough,ss)
Time Frame: Kel: 0 to 336 hours after the administration of the Cycle 7 infusion.
Population: Overall number of participants Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: l/h
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 55 | 61
l/h | 0.00236 (33.3) | 0.00240 (32.8)

13. Secondary Outcome: Volume of Distribution (Vd) of BEVZ92 and Avastin®
Description: Secondary PK endpoints included the Vd calculated at Cycle 7
Time Frame: Vd: 0 to 336 hours after the administration of the Cycle 7 infusion.
Population: In the Avastin arm there were several missing samples at the timepoint required for the specific PK parameter
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product).
Number analyzed (Participants) | 49 | 52
L | 4.06 (37.7) | 3.86 (39.4)

ADVERSE EVENTS:
Time Frame: Throughout the study (on day 1 of every cycle and 30 days after the end of study treatment). Adverse event data were collected from the beginning of the study at 29 Oct 2014 till last patient last visit in 10 Dec 2017 (Database lock point).
Description: Coded according to Medical Dictionary for Regulatory Activities (version 16.0), and graded on the basis of the US National Cancer Institute's Common Terminology for Adverse Events (version 4.0).
Arm/Group | Bevacizumab Biosimilar (BEVZ92) | Avastin® (Bevacizumab, Ref. Product)
All-Cause Mortality (participants affected / at risk) | 11/69 | 7/71
Serious Adverse Events (participants affected / at risk) | 19/69 | 21/71
Other Adverse Events (participants affected / at risk) | 66/69 | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Biosimilar (BEVZ92) (N=69) | Avastin® (Bevacizumab, Ref. Product) (N=71)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 5 (6) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Catheter site abscess (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Diarrhea infectious (Infections and infestations) | 1 (1) | 0 (0)
Pelvic Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (6)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) — Included in All-cause mortality
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Multi- organ failure (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) — Included in All-cause mortality
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Vena Cava Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Acute Kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Eye hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Cholecystis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Biosimilar (BEVZ92) (N=69) | Avastin® (Bevacizumab, Ref. Product) (N=71)
Diarrhea (Gastrointestinal disorders) | 34 | 41
Nausea (Gastrointestinal disorders) | 31 | 32
Vomiting (Gastrointestinal disorders) | 25 | 24
Constipation (Gastrointestinal disorders) | 9 | 19
Abdominal pain (Gastrointestinal disorders) | 6 | 18
Stomatitis (Gastrointestinal disorders) | 9 | 8
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5
Intestinal obstruction (Gastrointestinal disorders) | 5 | 1
Proctalgia (Gastrointestinal disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 22 | 21
Fatigue (General disorders) | 16 | 18
Pyrexia (General disorders) | 6 | 14
Mucosal inflammation (General disorders) | 7 | 6
Edema peripheral (General disorders) | 3 | 6
Neuropathy peripheral (Nervous system disorders) | 13 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 16
Paresthesia (Nervous system disorders) | 10 | 10
Headache (Nervous system disorders) | 7 | 10
Dysgeusia (Nervous system disorders) | 4 | 12
Dizziness (Nervous system disorders) | 4 | 4
Dysesthesia (Nervous system disorders) | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 23 | 26
Anemia (Blood and lymphatic system disorders) | 19 | 28
Leukopenia (Blood and lymphatic system disorders) | 14 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 13
Decreased appetite (Metabolism and nutrition disorders) | 19 | 20
Hypertriglyceridemia (Metabolism and nutrition disorders) | 11 | 17
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 10
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4
Urinary tract infection (Infections and infestations) | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 6
Influenza (Infections and infestations) | 6 | 5
Respiratory tract infection viral (Infections and infestations) | 4 | 3
Viral upper respiratory tract infection (Infections and infestations) | 4 | 1
Weight decreased (Investigations) | 16 | 12
Alanine aminotransferase increased (Investigations) | 8 | 9
Aspartate aminotransferase increased (Investigations) | 4 | 10
Blood creatinine increased (Investigations) | 2 | 6
Blood alkaline phosphatase increased (Investigations) | 2 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4
Hypertension (Vascular disorders) | 17 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Proteinuria (Renal and urinary disorders) | 7 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No